CLINICAL TRIAL: NCT06195423
Title: The Stop Osteoarthritis (SOAR) Hybrid Effectiveness-Implementation Type 1 Randomized Controlled Trial for Young People At-High-Risk of Early Onset Knee Osteoarthritis
Brief Title: Stopping OsteoARthritis After an ACL Tear
Acronym: SOAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Arthritis Research Centre of Canada (Other); The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Jackie Whittaker, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# H23-03544
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament Rupture; Osteoarthritis, Knee
Keywords: Randomized controlled trial; Post-traumatic osteoarthritis; Knee; Osteoarthritis prevention; Exercise; Rehabilitation
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Intervention Model Description: The proposed trial is a two-arm, assessor-blinded, superiority, hybrid effectiveness-implementation type 1 RCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop OsteoARthritis (SOAR) program (Experimental): Participants with a first-time ACL tear followed by reconstruction surgery randomized to the SOAR program group will complete a 6-month SOAR program (one-time Knee Camp, weekly home-based exercise therapy and physical activity with tracking, weekly 1:1 physiotherapist counseling sessions, and optional weekly group-based exercise classes) Consented trained physiotherapists will deliver the SOAR program throughout the study period to one or more SOAR program participants. Physiotherapists and SOAR participants will be randomly paired.
  Interventions: Behavioral: Stop OsteoARthritis (SOAR) program
- Living Well after ACLR (Active Comparator): Participants with a first-time ACL tear followed by reconstruction surgery randomized to the minimal control (Living Well after ACLR) group will complete a 6-month minimal intervention control program (educational video, workbook, activity tracking, and one 1:1 physiotherapist counseling session).
  Interventions: Behavioral: Living Well after ACLR program

INTERVENTIONS:
Behavioral: Stop OsteoARthritis (SOAR) program — The SOAR program is a 6-month, online-delivered (videoconferencing), PT-guided knee health program which consists of;
  1. Knee Camp: Includes interactive education, and 1:1 physiotherapy knee exam and counseling session to co-identify home-based exercise-therapy and physical activity goals to address participants' unique functional limitations. Participants are given a wrist-worn activity monitor to wear 24hours/day.
  2. Individualized Weekly Home-based Exercise-Therapy and Physical Activity Program: At home, participants work to meet their exercise-therapy and physical activity goals. Exercises and physical activity are tracked with an online form and the activity monitor. Participants can also attend an optional weekly group class.
  3. Weekly PT-guided Exercise-Therapy and Physical Activity Counselling: Each week, participants attend a 1:1 physiotherapist counseling session to modify exercise-therapy and physical activity goals.
  Other Names: SOAR
  Arms: Stop OsteoARthritis (SOAR) program
Behavioral: Living Well after ACLR program — Participants in the minimal intervention CONTROL group will receive access to a 30-minute educational video (knee anatomy, ACLR information, general exercise, physical activity, and goal-setting principles), a best practice workbook, one video-recorded virtual session with a physiotherapist (naïve to SOAR) who will explain the booklet and answer questions but not volunteer information beyond the video or booklet and the same wrist-worn activity tracker as the experimental group.
  Other Names: CONTROL
  Arms: Living Well after ACLR

SUMMARY:
By 2040, 25% of Canadians will have osteoarthritis, a disabling joint condition. Most people think osteoarthritis only affects older adults, but 50% of the 700,000 Canadian youth who hurt their knee playing sports annually will develop osteoarthritis by 40 years of age. These young people with old knees face knee pain and disability for much of their adult lives, interfering with parenting, work, and recreation. Yet, most do not know about osteoarthritis or how to reduce their risk.

In this clinical trial, people who have torn the Anterior Cruciate ligament in their knee and had reconstruction surgery 9-36 months previously will be randomized to receive either a 6-month virtual education and exercise therapy program called Stop OsteoARthritis (SOAR) or a minimal intervention control program. Researchers will test if those who received the SOAR program have larger gains in knee health, including pain, symptoms, function, and quality of life at 6, 12, and 24 months. Researchers will also use MRIs (baseline and 24 months) to assess how the SOAR program influences knee cartilage degeneration and its cost-effectiveness.

DETAILED DESCRIPTION:
PURPOSE: Assess the effectiveness, efficiency, and implementation of a 6-month evidence-informed, digital (online), education and exercise-therapy program (SOAR - Stop OsteoARthritis) versus a minimal intervention control for people aged 16-35 years at risk of early-onset knee osteoarthritis (OA) due to a first time Anterior Cruciate Ligament Reconstruction (ACLR).

OBJECTIVES:

Primary Effectiveness Objective: Assess if self-reported knee pain, symptoms, function, and QoL (average of the Knee injury and OA Outcome Score pain, other symptoms, function in sport and recreation, and quality of life subscale scores; KOOS4) of people at risk of knee OA who receive SOAR is superior to those receiving a minimal intervention CONTROL at 6 (primary end-point), 12, and 24 months.

Primary Efficiency Objective: Assess the incremental cost-utility ratio of SOAR compared CONTROL (6, 12, 24 months)

Primary Implementation Objective: Assess provider adoption of the SOAR program.

Secondary Effectiveness Objectives:

1. Assess if the perceived self-management of people at risk of knee OA who receive SOAR is superior to those receiving a minimal intervention CONTROL (6, 12, 24 months)
2. Assess if the percentage of SOAR group participants who achieve a Patient Acceptable Symptom State (PASS) for knee-related pain, other symptoms, function in daily living, function in sport and recreation, and quality of life is superior to CONTROL (6, 12, 24 months)
3. Assess if knee OA MRI features of SOAR group participants are superior to CONTROL (24 months)

Secondary Efficiency Objectives:

1. Describe the health resource use of SOAR and CONTROL participants (24 months)
2. Describe SOAR program delivery costs

Secondary Implementation Objectives:

1. Describe provider perceived barriers and facilitators of SOAR delivery
2. Describe participants' perceived barriers and facilitators of SOAR delivery
3. Describe features of physiotherapy (PT) counseling that promote self-management

Exploratory Effectiveness Objectives: Explore the superiority of SOAR to CONTROL on the following outcomes (at 6, 12, and 24 months);

1. Patient-specific function
2. Knee-related self-efficacy
3. Knee-related fear of movement and re-injury
4. Knee extensor strength
5. Knee flexor strength
6. Physical activity,
7. Health-related quality-of-life
8. Adiposity
9. Early cartilage degeneration (at 24 months only)

RESEARCH DESIGN:

The proposed trial is a two-arm, assessor-blinded, superiority, hybrid effectiveness-implementation type 1 randomized controlled trial with embedded cost-utility analyses and 1:1 interviews. This multi-focus design (effectiveness, implementation, efficacy) can accelerate research translation to real-world settings (Type 1: main focus-intervention effectiveness; secondary focus-understand implementation context). This design is appropriate as we have shown feasibility and indirect evidence of SOAR effect, the intervention is minimal risk, and there are no fully powered superiority trials to inform non-inferiority or equivalence designs.

The nature of the interventions do not allow for full blinding (physiotherapists cannot be blinded to treatment). We will employ proven methods from our proof-of-concept RCT to reduce allocation (online randomization module with schedule prepared by an arms-length statistician) and confirmation bias (outcome assessors and data analysts will be blinded to allocation).

STATISTICAL ANALYSES:

Primary analyses will be intent-to-treat (by randomization). Data missing more than 5% will be imputed using multiple imputations by chained equations to avoid bias. To ensure best practice, all outcome and demographic/prognostic variables will be included in imputation equations.

Demographics: Descriptive statistics will be calculated for demographic and potentially prognostic variables (time since injury and ACLR, concomitant injury, ACLR rehabilitation, graft type, reinjury, co-intervention, SES) and observed differences considered or controlled for when interpreting findings.

Effectiveness: SOAR superiority will be assessed with a generalized linear mixed regression model (GLMM) for the primary outcome (KOOS4 at 6 months) adjusted for baseline measure, time since ACLR, and sex. Adjusting for continuous time since ACLR versus stratifying improves power. Similar GLMMs will assess SOAR superiority for continuous secondary (PIH) and exploratory (knee extensor strength, adiposity, physical activity) outcomes at stated time points. Mixed effect logistic regression models (adjusted for the same variables as GLMMs) will assess SOAR superiority for binary secondary outcomes (MRI lesion worsening, achieving PASS) at stated time points. Analyses will yield valid results under the missing at random (MAR) assumption. The robustness of estimates to potential MAR assumption violations will be assessed with state-of-art methods.

Sex/Gender: To explore the effect of gender identity (women, man, gender-diverse) and sex (female, male, intersex) on outcome variables and intervention effect, all outcomes will be described by treatment group stratified by gender (KOOS4, Partner in Health Scale, cost-utility, physical activity, quality of life) or sex (MRI, knee extensor strength, adiposity) at all time points. We will estimate GLMMs and report intervention effect estimates stratified by sex (female, male) or gender (woman, man) as exploratory analyses to inform future studies. As 6% of our preliminary proof-of-concept randomized controlled trial participants identified gender diverse, descriptive statistics will also explore differences by cis and diverse gender.

Implementation: The % of physiotherapists achieving ≥85% on the fidelity checklist and checklist items with ≤70% fidelity will be reported. Provider and participants' responses to survey questions asking about barriers and facilitators of SOAR implementation will be summarized. Interview recordings related to identifying features of participant-provider interactions that facilitate self-management will be transcribed and de-identified. Data will be coded using a constant comparative approach, and categories will be developed by comparing and identifying meaningful patterns across codes. High-order themes will elucidate the relationship between categories. We will look for uniqueness by gender and, if found, reanalyze the data with a gender lens. Analysis trustworthiness and credibility will be fostered through data immersion, memoing, reflexive journaling, and team discussions. An audit of analytic decisions will be kept.

Efficiency outcome: Incremental cost-utility ratio will be estimated as (Cost_SOAR - Cost_CONTROL) ⁄(∆QALY_SOAR - ∆QALY_CONTROL) for the intervention and 6-month post-intervention period using nested imputation and nonparametric bootstrapping to model uncertainty around cost and QALY estimates. The contribution of each cost item to total healthcare resource use will be described by group, gender, and compliance (full, partial).

ELIGIBILITY:
Inclusion Criteria:

* Currently live in British Columbia, Canada
* 16-35 years of age (inclusive)
* 9-36-months past a first-time ACLR performed ≤12-months of first-time ACL tear
* Currently not receiving knee care from a health or fitness provider and have no scheduled surgical procedures (any part of the body) that would interfere with exercise during the study.
* Score below a KOOS4 PASS (<79 points)
* Have daily access to an email address and a computer with internet
* Are willing to wear an activity tracker during the study

Exclusion Criteria:

* Inability to communicate in English
* No medical attention (healthcare provider) time-loss (missed physical activity, sport or work ≥2 occasions) injury to the ACLR knee before the ACL tear
* Previous physician diagnosis of index knee osteoarthritis
* Inflammatory arthritis or other systemic condition
* Lower limb injury, surgery, or intra-articular injection in the past 6-months
* Current pregnancy
* MRI contraindications (i.e., Weight over 400 lbs (MRI machine limit); Pacemaker or any other implanted medical device (i.e., wires, defibrillator, artificial heart valve, an electronic device like a drug infusion pump, electrical stimulator for nerves or bones, coil, catheter, or filter in any blood vessel, ear or eye implant, or stainless steel intrauterine device (IUD); Brain or ferromagnetic aneurysm clip; any other metallic prostheses or shrapnel, bullets, or other metal fragments; injury where a piece of metal lodged in the eye or orbit, or; surgery, medical procedure or tattoos (including tattooed eyeliner) in the last 6 weeks).

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported knee-related pain, symptoms, function in sport and quality of life over 6 months (effectiveness outcome) (ACL tear participants) | Change from baseline KOOS score at 6 months (ACL tear participants)
  Patient partners identify pain, function and quality of life, which can be impaired up to 10-years post-ACLR, as priority outcomes. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a valid and reliable patient-reported outcome measure (PROM) with sub-scales for knee pain (9-items), other symptoms (7-items), function in daily living (ADL; 17-items), function in sport/recreation (5-items), and quality of life (4-items) across injury and OA populations. Each subscale item is scored on a 5-point scale and individual subscale items summed and transformed to a 0-100 scale with higher scores indicating better outcome. The KOOS4 which is an average of 4 sub-scales (excluding ADL) is a recommended and accepted primary outcome for ACLR RCTs and was responsive in our proof of concept RCT.
Incremental cost-utility ratio over 6 months (efficiency outcome) | Incremental cost-utility ratio at 6 months
  To assess SOARs value for money (health systems perspective) we will estimate the incremental cost/mean change in Quality-Adjusted Life Years (QALY) gained by SOAR versus CONTROL at 6 months. Costs will be estimated with the Health Resource Utilization questionnaire (HRU) as the study population often uses resources not captured in administrative data and evidence of good agreement between administrative and prospectively collected HRU data. The HRU captures provider visits, hospital admissions, lab and diagnostic tests and medication use. QALYs will be estimated from health-related quality of life (EQ-5D-5L) using area under the curve analysis. The EQ-5D-5L is widely used for cost-utility analyses in OA, and assesses 5 levels across 5 health domains to produce a health state profile using Canadian conversion tariffs.
Provider adoption of SOAR over 6 months (implementation outcome) (physiotherapist participants) | Percent fidelity at 6 months (physiotherapist participants)
  A 40-item fidelity checklist, refined in our proof-of-concept RCT, will be applied to all video-recorded 1:1 counseling sessions for 4 participants per PT, and the median % fidelity for each PT and checklist item reported. Items reaching ≤70% will be identified and inform the development of PT training modules to facilitate future evaluation and implementation.

SECONDARY OUTCOMES:
Patient Acceptable Symptom State over 6 months (ACL tear participants) | Change from baseline patient acceptable symptom state score at 6 months (ACL tear participants)
  To help interpret the clinical relevance of the KOOS4, the percentage of participants in both study groups to reach KOOS4 and KOOS sub-scale Patient Acceptable Symptom State (PASS) scores (KOOS4 79; pain 89; symptoms 83; ADL 95, sport 72; QoL 73) will be reported.
Self-reported perceived self-management over 6 months (ACL tear participants) | Change from baseline self-reported perceived self-management at 6 months (ACL tear participants)
  The 12 item Partner in Health Scale will be used to measure perceived self-management (active involvement to self-manage a chronic condition). Each item is scored on a 0-9 point Likert scale. Scores on individual items are summed to produce a total score ranging between 0 and 96, with 0 representing no perceived self-management and 96 representing full perceived self-management. The total time for this questionnaire is 3 minutes. The Partner in Health Scale is valid and reliable across numerous chronic conditions.
Osteoarthritis MRI features over 24 months (ACL tear participants) | Change from baseline MRI at 24 months (ACL tear participants)
  MRI features of OA (cartilage defect, bone marrow lesions) are important for early disease staging and common after ACLR. The impact of exercise on these outcomes post-ACLR is unknown. The valid semi-quantitative MRI OA knee score (MOAKS) will be applied to 3D proton-density (PD) gradient MRI sequences (3T scanner, Philips Elition, 8-channel knee coil). Positioning aids will immobilize the knee to ensure consistent scans. Radiology fellows will conduct MOAKS ratings blinded to group allocation. OA feature worsening will be defined as an increase in the size of the lesion using established methods.
Health resource use costs over 24 months | Health resource use costs over 24 months
  Monthly health resource use costs (HRU) will be reported over the 24-month study period.
Intervention delivery costs over 6 months | Intervention delivery costs over 6 months
  The cost to deliver the SOAR and CONTROL (Living Well with ACLR) interventions will be tracked and reported.
Participant perceived barriers and facilitators of program delivery over 6 months (ACL tear participants) | Follow-up surveys will take place at 6 months (ACL tear participants)
  On completion of the intervention, participants will receive a follow-up survey which will include questions to capture information about their perceived barriers and facilitators of program delivery, and therapeutic alliance with their PT (Consultation and Relational Empathy measure (CARE)).
Provider perceived barriers and facilitators of program delivery over 6 months (physiotherapist participants) | Follow-up surveys will take place at 6 months (physiotherapist participants)
  After PT's are done delivering the SOAR program they will receive a follow-up survey including questions to capture information about their perceived barriers and facilitators of SOAR program delivery, SOAR and BAP training, confidence in BAP, SMART goal setting, shared decision making, virtual PT delivery, and perceived impacts on patient and clinic flow.
Features of PT counselling that promote self-management over 6 months (ACL tear participants) | 1:1 interviews will be conducted at 6 months (ACL tear participants)
  Semi-structured 1:1 interviews will be conducted with a purposive maximum variation sample (gender, age, adherence, time since injury) of 15-20 participants. Using video-cued narrative reflection, participants will self-select meaningful exchanges with their PT that promoted self-management while viewing a Knee Camp recording and a random weekly counselling session. Participants will be able to pause and rewind the recording to identify, and elaborate on significant moments. A definition of self-management and context-specific examples will be provided. Probe and prompts will provide elaboration. Field notes will be taken, and interviews recorded. Ongoing analyses will inform sampling, and data collection will cease when no new themes are identified. Video-recorded healthcare interactions are acceptable and provide valuable practice insights. Video-cued interviews yield rich data as participants simultaneously identify, engage and reflect on their lived experience.

OTHER OUTCOMES:
Self-reported knee-related pain, symptoms, function in sport and quality of life over 12 months (ACL tear participants) | Change from baseline KOOS score at 12 months (ACL tear participants)
  Patient partners identify pain, function and quality of life, which can be impaired up to 10-years post-ACLR, as priority outcomes. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a valid and reliable patient-reported outcome measure (PROM) with sub-scales for knee pain (9-items), other symptoms (7-items), function in daily living (ADL; 17-items), function in sport/recreation (5-items), and quality of life (4-items) across injury and OA populations. Each subscale item is scored on a 5-point scale and individual subscale items summed and transformed to a 0-100 scale with higher scores indicating better outcome. The KOOS4 which is an average of 4 sub-scales (excluding ADL) is a recommended and accepted primary outcome for ACLR RCTs and was responsive in our proof of concept RCT.
Self-reported knee-related pain, symptoms, function in sport and quality of life over 24 months (ACL tear participants) | Change from baseline KOOS score at 24 months (ACL tear participants)
  Patient partners identify pain, function and quality of life, which can be impaired up to 10-years post-ACLR, as priority outcomes. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a valid and reliable patient-reported outcome measure (PROM) with sub-scales for knee pain (9-items), other symptoms (7-items), function in daily living (ADL; 17-items), function in sport/recreation (5-items), and quality of life (4-items) across injury and OA populations. Each subscale item is scored on a 5-point scale and individual subscale items summed and transformed to a 0-100 scale with higher scores indicating better outcome. The KOOS4 which is an average of 4 sub-scales (excluding ADL) is a recommended and accepted primary outcome for ACLR RCTs and was responsive in our proof of concept RCT.
Incremental cost-utility ratio over 12 months | Incremental cost-utility ratio at 12 months
  To assess SOARs value for money (health systems perspective) we will estimate the incremental cost/mean change in Quality-Adjusted Life Years (QALY) gained by SOAR versus CONTROL at 12 months. Costs will be estimated with the Health Resource Utilization questionnaire (HRU) as the study population often uses resources not captured in administrative data and evidence of good agreement between administrative and prospectively collected HRU data. The HRU captures provider visits, hospital admissions, lab and diagnostic tests and medication use. QALYs will be estimated from health-related quality of life (EQ-5D-5L) using area under the curve analysis. The EQ-5D-5L is widely used for cost-utility analyses in OA, and assesses 5 levels across 5 health domains to produce a health state profile using Canadian conversion tariffs.
Incremental cost-utility ratio over 24 months | Incremental cost-utility ratio at 24 months
  To assess SOARs value for money (health systems perspective) we will estimate the incremental cost/mean change in Quality-Adjusted Life Years (QALY) gained by SOAR versus CONTROL at 24 months. Costs will be estimated with the Health Resource Utilization questionnaire (HRU) as the study population often uses resources not captured in administrative data and evidence of good agreement between administrative and prospectively collected HRU data. The HRU captures provider visits, hospital admissions, lab and diagnostic tests and medication use. QALYs will be estimated from health-related quality of life (EQ-5D-5L) using area under the curve analysis. The EQ-5D-5L is widely used for cost-utility analyses in OA, and assesses 5 levels across 5 health domains to produce a health state profile using Canadian conversion tariffs.
Patient Acceptable Symptom State over 12 months (ACL tear participants) | Change from baseline Patient Acceptable Symptom State score at 12 months (ACL tear participants)
  To help interpret the clinical relevance of the KOOS4, the percentage of participants in both study groups to reach KOOS4 and KOOS sub-scale Patient Acceptable Symptom State (PASS) scores (KOOS4 79; pain 89; symptoms 83; ADL 95, sport 72; QoL 73) will be reported.
Patient Acceptable Symptom State over 24 months (ACL tear participants) | Change from baseline Patient Acceptable Symptom State score at 24 months (ACL tear participants)
  To help interpret the clinical relevance of the KOOS4, the percentage of participants in both study groups to reach KOOS4 and KOOS sub-scale Patient Acceptable Symptom State (PASS) scores (KOOS4 79; pain 89; symptoms 83; ADL 95, sport 72; QoL 73) will be reported.
Self-reported perceived self-management over 12 months (ACL tear participants) | Change from baseline self-reported perceived self-management at 12 months (ACL tear participants)
  The 12 item Partner in Health Scale will be used to measure perceived self-management (active involvement to self-manage a chronic condition). Each item is scored on a 0-9 point Likert scale. Scores on individual items are summed to produce a total score ranging between 0 and 96, with 0 representing no perceived self-management and 96 representing full perceived self-management. The total time for this questionnaire is 3 minutes. The Partner in Health Scale is valid and reliable across numerous chronic conditions.
Perceived self-management over 24 months (ACL tear participants) | Change from baseline self-reported perceived self-management at 24 months (ACL tear participants)
  The 12 item Partner in Health Scale will be used to measure perceived self-management (active involvement to self-manage a chronic condition). Each item is scored on a 0-9 point Likert scale. Scores on individual items are summed to produce a total score ranging between 0 and 96, with 0 representing no perceived self-management and 96 representing full perceived self-management. The total time for this questionnaire is 3 minutes. The Partner in Health Scale is valid and reliable across numerous chronic conditions.
Self-reported function over 6 months (ACL tear participants) | Change from baseline self-reported function at 6 months (ACL tear participants)
  The 3 item Patient Specific Functional Scale will be used to identify, quantify and assess changes in functional limitations that are most relevant to participants. This scale prompts participants to identify three activities important to them and rate their ability to perform each activity on a 10-point numerical rating scale. Individual scale scores are summed and transformed to a 0-100 scale with higher scores indicating better outcomes. The total time for this questionnaire is 3 minutes. The Patient-Specific Functional Scale is valid and reliable for use in persons with a knee injury.
Self-reported function over 12 months (ACL tear participants) | Change from baseline self-reported function at 12 months (ACL tear participants)
  The 3 item Patient Specific Functional Scale will be used to identify, quantify and assess changes in functional limitations that are most relevant to participants. This scale prompts participants to identify three activities important to them and rate their ability to perform each activity on a 10-point numerical rating scale. Individual scale scores are summed and transformed to a 0-100 scale with higher scores indicating better outcomes. The total time for this questionnaire is 3 minutes. The Patient-Specific Functional Scale is valid and reliable for use in persons with a knee injury.
Self-reported function over 24 months (ACL tear participants) | Change from baseline self-reported function at 24 months (ACL tear participants)
  The 3 item Patient Specific Functional Scale will be used to identify, quantify and assess changes in functional limitations that are most relevant to participants. This scale prompts participants to identify three activities important to them and rate their ability to perform each activity on a 10-point numerical rating scale. Individual scale scores are summed and transformed to a 0-100 scale with higher scores indicating better outcomes. The total time for this questionnaire is 3 minutes. The Patient-Specific Functional Scale is valid and reliable for use in persons with a knee injury.
Self-reported knee-specific self-efficacy over 6 months (ACL tear participants) | Change from baseline self-reported knee-specific self-efficacy at 6 months (ACL tear participants)
  Self-efficacy, or one's belief in their own ability to organize and execute the actions required to manage a prospective situation, can predict health behaviours including exercise participation. The KSES is a valid and reliable measure of knee-specific self-efficacy in people with a sport-related knee injury in the previous 5-years. The KSES consists of 22 items organized into 2 sub-scales (present and future self-efficacy). Each item is scored on an 0-10-point Likert scale, with 0 indicating no confidence and 10 indicating full confidence. Individual item scores are summed to produce a total score. Higher scores indicate higher levels of self-efficacy.
Self-reported knee-specific self-efficacy over 12 months (ACL tear participants) | Change from baseline self-reported knee-specific self-efficacy at 12 months (ACL tear participants)
  Self-efficacy, or one's belief in their own ability to organize and execute the actions required to manage a prospective situation, can predict health behaviours including exercise participation. The KSES is a valid and reliable measure of knee-specific self-efficacy in people with a sport-related knee injury in the previous 5-years. The KSES consists of 22 items organized into 2 sub-scales (present and future self-efficacy). Each item is scored on an 0-10-point Likert scale, with 0 indicating no confidence and 10 indicating full confidence. Individual item scores are summed to produce a total score. Higher scores indicate higher levels of self-efficacy.
Self-reported knee-specific self-efficacy over 24 months (ACL tear participants) | Change from baseline self-reported knee-specific self-efficacy at 24 months (ACL tear participants)
  Self-efficacy, or one's belief in their own ability to organize and execute the actions required to manage a prospective situation, can predict health behaviours including exercise participation. The KSES is a valid and reliable measure of knee-specific self-efficacy in people with a sport-related knee injury in the previous 5-years. The KSES consists of 22 items organized into 2 sub-scales (present and future self-efficacy). Each item is scored on an 0-10-point Likert scale, with 0 indicating no confidence and 10 indicating full confidence. Individual item scores are summed to produce a total score. Higher scores indicate higher levels of self-efficacy.
Self-reported fear of movement and re-injury over 6 months (ACL tear participants) | Change from baseline self-reported fear of movement and re-injury at 6 months (ACL tear participants)
  The 11 item Tampa Scale of Kinesiophobia will be used to measure self-reported fear of movement and re-injury. Each item is scored on a 0-4 point Likert-scale, with 0 indicating no fear of movement and 4 indicating greater fear of movement. The item scores are summed to produce a total score ranging between 0 and 44, with higher values indicating a higher degree of fear of movement. The total time for this questionnaire is 3 minutes. The Tampa Scale of Kinesiophobia has evidence of known-group validity (scores discriminated between athletes who returned and did not return to pre-injury sports participation level after knee trauma).
Self-reported fear of movement and re-injury over 12 months (ACL tear participants) | Change from baseline self-reported fear of movement and re-injury at 12 months (ACL tear participants)
  The 11 item Tampa Scale of Kinesiophobia will be used to measure self-reported fear of movement and re-injury. Each item is scored on a 0-4 point Likert-scale, with 0 indicating no fear of movement and 4 indicating greater fear of movement. The item scores are summed to produce a total score ranging between 0 and 44, with higher values indicating a higher degree of fear of movement. The total time for this questionnaire is 3 minutes. The Tampa Scale of Kinesiophobia has evidence of known-group validity (scores discriminated between athletes who returned and did not return to pre-injury sports participation level after knee trauma).
Self-reported fear of movement and re-injury over 24 months (ACL tear participants) | Change from baseline self-reported fear of movement and re-injury at 24 months (ACL tear participants)
  The 11 item Tampa Scale of Kinesiophobia will be used to measure self-reported fear of movement and re-injury. Each item is scored on a 0-4 point Likert-scale, with 0 indicating no fear of movement and 4 indicating greater fear of movement. The item scores are summed to produce a total score ranging between 0 and 44, with higher values indicating a higher degree of fear of movement. The total time for this questionnaire is 3 minutes. The Tampa Scale of Kinesiophobia has evidence of known-group validity (scores discriminated between athletes who returned and did not return to pre-injury sports participation level after knee trauma).
Change in Knee Extension Power over 6 months (ACL tear participants) | Change from baseline knee extensor muscle power at 6 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee extension power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to straighten their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Extension Power over 12 months (ACL tear participants) | Change from baseline knee extensor muscle power at 12 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee extension power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to straighten their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Extension Power over 24 months (ACL tear participants) | Change from baseline knee extensor muscle power at 24 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee extension power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to straighten their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Flexion Power over 6 months (ACL tear participants) | Change from baseline knee extensor muscle power at 6 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee flexion power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to bend their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Flexion Power over 12 months (ACL tear participants) | Change from baseline knee extensor muscle power at 12 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee flexion power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to bend their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Flexion Power over 24 months (ACL tear participants) | Change from baseline knee extensor muscle power at 24 months (ACL tear participants)
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee flexion power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to bend their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Daily Average Moderate to Vigorous Physical Activity over 6 months (ACL tear participants) | Change from baseline daily average moderate to vigorous physical activity at 6 months (ACL tear participants)
  A small, lightweight hip worn wearable triaxial accelerometer (ActiGraph GT3X®) will be used to assess physical activity. Participants will be asked to wear this device (attached via an elastic belt around their waist), for a period of 7 consecutive days removing only for bathing/swimming activities. The average number of 10-minute moderate-to-vigorous physical activity bouts over the 7-day period will be calculated. Accelerometry is a valid measure of physical activity in youth and young adult populations.
Change in Daily Average Moderate to Vigorous Physical Activity over 12 months (ACL tear participants) | Change from baseline daily average moderate to vigorous physical activity at 12 months (ACL tear participants)
  A small, lightweight hip worn wearable triaxial accelerometer (ActiGraph GT3X®) will be used to assess physical activity. Participants will be asked to wear this device (attached via an elastic belt around their waist), for a period of 7 consecutive days removing only for bathing/swimming activities. The average number of 10-minute moderate-to-vigorous physical activity bouts over the 7-day period will be calculated. Accelerometry is a valid measure of physical activity in youth and young adult populations.
Change in Daily Average Moderate to Vigorous Physical Activity over 24 months (ACL tear participants) | Change from baseline daily average moderate to vigorous physical activity at 24 months (ACL tear participants)
  A small, lightweight hip worn wearable triaxial accelerometer (ActiGraph GT3X®) will be used to assess physical activity. Participants will be asked to wear this device (attached via an elastic belt around their waist), for a period of 7 consecutive days removing only for bathing/swimming activities. The average number of 10-minute moderate-to-vigorous physical activity bouts over the 7-day period will be calculated. Accelerometry is a valid measure of physical activity in youth and young adult populations.
Change in Self-Reported Physical Activity over 6 months (ACL tear participants) | Change from baseline self-reported physical activity at 6 months (ACL tear participants)
  The 4 item Godin Leisure Time Questionnaire will be used to measure self-reported physical activity. Using the number of 15-minute bouts of mild, moderate, and strenuous physical activity a participant engages in over a typical seven-day period weekly metabolic equivalents of physical activity are calculated. The total time for this questionnaire is 1 minute. The Godin Leisure Time Questionnaire has been validated to assess physical activity.
Change in Self-Reported Physical Activity over 12 months (ACL tear participants) | Change from baseline self-reported physical activity at 12 months (ACL tear participants)
  The 4 item Godin Leisure Time Questionnaire will be used to measure self-reported physical activity. Using the number of 15-minute bouts of mild, moderate, and strenuous physical activity a participant engages in over a typical seven-day period weekly metabolic equivalents of physical activity are calculated. The total time for this questionnaire is 1 minute. The Godin Leisure Time Questionnaire has been validated to assess physical activity.
Change in Self-Reported Physical Activity over 24 months (ACL tear participants) | Change from baseline self-reported physical activity at 24 months (ACL tear participants)
  The 4 item Godin Leisure Time Questionnaire will be used to measure self-reported physical activity. Using the number of 15-minute bouts of mild, moderate, and strenuous physical activity a participant engages in over a typical seven-day period weekly metabolic equivalents of physical activity are calculated. The total time for this questionnaire is 1 minute. The Godin Leisure Time Questionnaire has been validated to assess physical activity.
Change in Health-Related Quality of Life over 6 months (ACL tear participants) | Change from baseline health-related quality of life at 6 months (ACL tear participants)
  The EQ-5D-5L is a simple, reliable self-report instrument designed to assess generic health for clinical and economic appraisal across multiple countries and conditions (see attachment 16-EQ-5D-5L). The EQ-5D-5L provides information about 5 levels of problems across 5 health domains (anxiety/depression, pain/discomfort, mobility, self-care, usual activities), and a 0-to-100 visual analogue scale rating for self-related health (EQ-5D-5Lindex). EQ-5D-5Lindex values will be reported at each time point.
Change in Health-Related Quality of Life over 12 months (ACL tear participants) | Change from baseline health-related quality of life at 12 months (ACL tear participants)
  The EQ-5D-5L is a simple, reliable self-report instrument designed to assess generic health for clinical and economic appraisal across multiple countries and conditions (see attachment 16-EQ-5D-5L). The EQ-5D-5L provides information about 5 levels of problems across 5 health domains (anxiety/depression, pain/discomfort, mobility, self-care, usual activities), and a 0-to-100 visual analogue scale rating for self-related health (EQ-5D-5Lindex). EQ-5D-5Lindex values will be reported at each time point.
Change in Health-Related Quality of Life over 24 months (ACL tear participants) | Change from baseline health-related quality of life at 24 months (ACL tear participants)
  The EQ-5D-5L is a simple, reliable self-report instrument designed to assess generic health for clinical and economic appraisal across multiple countries and conditions (see attachment 16-EQ-5D-5L). The EQ-5D-5L provides information about 5 levels of problems across 5 health domains (anxiety/depression, pain/discomfort, mobility, self-care, usual activities), and a 0-to-100 visual analogue scale rating for self-related health (EQ-5D-5Lindex). EQ-5D-5Lindex values will be reported at each time point.
Change in Fat Mass Index over 6 months (ACL tear participants) | Change from baseline fat mass index at 6 months (ACL tear participants)
  Fat mass index (kg/m2) will be measured with Bioelectrical Impedance (Tanita Body Composition Analyzer, Model TBF-300A, Tanita Inc., USA). Participants will stand barefoot on the bioelectrical impedance platform during which the resistance to the flow of this single, high frequency alternating electrical current (500 A at 50 kHz) will be measured. Bioelectrical Impedance is a feasible method for assessing and tracking body composition in clinical settings and has been shown to be valid and reliable in child, youth, and adult populations. This test will take 5 minutes to complete. The device will be calibrated prior to each scan (according to the manufacturer's protocol).
Change in Fat Mass Index over 12 months (ACL tear participants) | Change from baseline fat mass index at 12 months (ACL tear participants)
  Fat mass index (kg/m2) will be measured with Bioelectrical Impedance (Tanita Body Composition Analyzer, Model TBF-300A, Tanita Inc., USA). Participants will stand barefoot on the bioelectrical impedance platform during which the resistance to the flow of this single, high frequency alternating electrical current (500 A at 50 kHz) will be measured. Bioelectrical Impedance is a feasible method for assessing and tracking body composition in clinical settings and has been shown to be valid and reliable in child, youth, and adult populations. This test will take 5 minutes to complete. The device will be calibrated prior to each scan (according to the manufacturer's protocol).
Change in Fat Mass Index over 24 months (ACL tear participants) | Change from baseline fat mass index at 24 months (ACL tear participants)
  Fat mass index (kg/m2) will be measured with Bioelectrical Impedance (Tanita Body Composition Analyzer, Model TBF-300A, Tanita Inc., USA). Participants will stand barefoot on the bioelectrical impedance platform during which the resistance to the flow of this single, high frequency alternating electrical current (500 A at 50 kHz) will be measured. Bioelectrical Impedance is a feasible method for assessing and tracking body composition in clinical settings and has been shown to be valid and reliable in child, youth, and adult populations. This test will take 5 minutes to complete. The device will be calibrated prior to each scan (according to the manufacturer's protocol).
Change in Knee Cartilage Health over 24 months (ACL tear participants) | Change from baseline knee cartilage health at 24 months (ACL tear participants)
  Preliminary research links exercise-therapy to better knee cartilage health in people at risk of post-traumatic OA (post-meniscectomy) and early atraumatic OA up to 12-months. We will provide further insight over 24-months by quantifying changes in cartilage T2 relaxation times (sagittal multi-echo-spin-echo pulse sequences;12 echos) which are widely used as a marker of early degeneration. An senior imaging scientist will segment the cartilage manually and calculate average T2 for femoral, tibial and patellar cartilage plates.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie L Whittaker, BScPT, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Arthritis Research Canada, Vancouver, British Columbia
  - Sea to Sky Orthopaedics, Whistler, British Columbia

REFERENCES:
- [Background] Bombardier C, Hawker G, Mosher D. The Impact of Arthritis in Canada: Today and Over the Next 30 Years. Arthritis Alliance of Canada. Fall 2011.
- [Background] Ackerman IN, Bohensky MA, Zomer E, Tacey M, Gorelik A, Brand CA, de Steiger R. The projected burden of primary total knee and hip replacement for osteoarthritis in Australia to the year 2030. BMC Musculoskelet Disord. 2019 Feb 23;20(1):90. doi: 10.1186/s12891-019-2411-9. PMID 30797228
- [Background] Sharif B, Kopec JA, Wong H, Anis AH. Distribution and Drivers of Average Direct Cost of Osteoarthritis in Canada From 2003 to 2010. Arthritis Care Res (Hoboken). 2017 Feb;69(2):243-251. doi: 10.1002/acr.22933. PMID 27159532
- [Background] Hunter DJ, Schofield D, Callander E. The individual and socioeconomic impact of osteoarthritis. Nat Rev Rheumatol. 2014 Jul;10(7):437-41. doi: 10.1038/nrrheum.2014.44. Epub 2014 Mar 25. PMID 24662640
- [Background] Sharif B, Garner R, Sanmartin C, Flanagan WM, Hennessy D, Marshall DA. Risk of work loss due to illness or disability in patients with osteoarthritis: a population-based cohort study. Rheumatology (Oxford). 2016 May;55(5):861-8. doi: 10.1093/rheumatology/kev428. Epub 2016 Jan 11. PMID 26759430
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Tugwell P, Bennett KJ, Sackett DL, Haynes RB. The measurement iterative loop: a framework for the critical appraisal of need, benefits and costs of health interventions. J Chronic Dis. 1985;38(4):339-51. doi: 10.1016/0021-9681(85)90080-3. PMID 3923014
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Runhaar J, Schiphof D, van Meer B, Reijman M, Bierma-Zeinstra SM, Oei EH. How to define subregional osteoarthritis progression using semi-quantitative MRI osteoarthritis knee score (MOAKS). Osteoarthritis Cartilage. 2014 Oct;22(10):1533-6. doi: 10.1016/j.joca.2014.06.022. PMID 25278062
- [Background] Hunter DJ, Guermazi A, Lo GH, Grainger AJ, Conaghan PG, Boudreau RM, Roemer FW. Evolution of semi-quantitative whole joint assessment of knee OA: MOAKS (MRI Osteoarthritis Knee Score). Osteoarthritis Cartilage. 2011 Aug;19(8):990-1002. doi: 10.1016/j.joca.2011.05.004. Epub 2011 May 23. PMID 21645627
- [Background] Truong LK, Mosewich AD, Miciak M, Pajkic A, Silvester-Lee T, Li LC, Whittaker JL. "I feel I'm leading the charge." Experiences of a virtual physiotherapist-guided knee health program for persons at-risk of osteoarthritis after a sport-related knee injury. Osteoarthr Cartil Open. 2022 Dec 27;5(1):100333. doi: 10.1016/j.ocarto.2022.100333. eCollection 2023 Mar. PMID 36685259
- [Background] Whittaker JL, Truong LK, Silvester-Lee T, Losciale JM, Miciak M, Pajkic A, Le CY, Hoens AM, Mosewich AD, Hunt MA, Li LC, Roos EM. Feasibility of the SOAR (Stop OsteoARthritis) program. Osteoarthr Cartil Open. 2022 Jan 28;4(1):100239. doi: 10.1016/j.ocarto.2022.100239. eCollection 2022 Mar. PMID 36474472
- [Background] Whittaker JL, Truong LK, Losciale JM, Silvester-Lee T, Miciak M, Pajkic A, Le CY, Hoens AM, Mosewich A, Hunt MA, Li LC, Roos EM. Efficacy of the SOAR knee health program: protocol for a two-arm stepped-wedge randomized delayed-controlled trial. BMC Musculoskelet Disord. 2022 Jan 25;23(1):85. doi: 10.1186/s12891-022-05019-z. PMID 35078446
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Culvenor AG, West TJ, Bruder AM, Scholes MJ, Barton CJ, Roos EM, Oei E, McPhail SM, Souza RB, Lee J, Patterson BE, Girdwood MA, Couch JL, Crossley KM. SUpervised exercise-therapy and Patient Education Rehabilitation (SUPER) versus minimal intervention for young adults at risk of knee osteoarthritis after ACL reconstruction: SUPER-Knee randomised controlled trial protocol. BMJ Open. 2023 Jan 18;13(1):e068279. doi: 10.1136/bmjopen-2022-068279. PMID 36657757
- [Background] Roos EM, Boyle E, Frobell RB, Lohmander LS, Ingelsrud LH. It is good to feel better, but better to feel good: whether a patient finds treatment 'successful' or not depends on the questions researchers ask. Br J Sports Med. 2019 Dec;53(23):1474-1478. doi: 10.1136/bjsports-2018-100260. Epub 2019 May 9. PMID 31072841
- [Background] Whittaker JL, Toomey CM, Nettel-Aguirre A, Jaremko JL, Doyle-Baker PK, Woodhouse LJ, Emery CA. Health-related Outcomes after a Youth Sport-related Knee Injury. Med Sci Sports Exerc. 2019 Feb;51(2):255-263. doi: 10.1249/MSS.0000000000001787. PMID 30239493
- [Background] Whittaker JL, Culvenor AG, Juhl CB, Berg B, Bricca A, Filbay SR, Holm P, Macri E, Urhausen AP, Ardern CL, Bruder AM, Bullock GS, Ezzat AM, Girdwood M, Haberfield M, Hughes M, Ingelsrud LH, Khan KM, Le CY, Losciale JM, Lundberg M, Miciak M, Oiestad BE, Patterson B, Raisanen AM, Skou ST, Thorlund JB, Toomey C, Truong LK, Meer BLV, West TJ, Young JJ, Lohmander LS, Emery C, Risberg MA, van Middelkoop M, Roos EM, Crossley KM. OPTIKNEE 2022: consensus recommendations to optimise knee health after traumatic knee injury to prevent osteoarthritis. Br J Sports Med. 2022 Dec;56(24):1393-1405. doi: 10.1136/bjsports-2022-106299. Epub 2022 Nov 15. PMID 36379676
- [Background] Smith D, Harvey P, Lawn S, Harris M, Battersby M. Measuring chronic condition self-management in an Australian community: factor structure of the revised Partners in Health (PIH) scale. Qual Life Res. 2017 Jan;26(1):149-159. doi: 10.1007/s11136-016-1368-5. Epub 2016 Jul 18. PMID 27432251
- [Background] Chatman AB, Hyams SP, Neel JM, Binkley JM, Stratford PW, Schomberg A, Stabler M. The Patient-Specific Functional Scale: measurement properties in patients with knee dysfunction. Phys Ther. 1997 Aug;77(8):820-9. doi: 10.1093/ptj/77.8.820. PMID 9256870
- [Background] Thomee P, Wahrborg P, Borjesson M, Thomee R, Eriksson BI, Karlsson J. Self-efficacy, symptoms and physical activity in patients with an anterior cruciate ligament injury: a prospective study. Scand J Med Sci Sports. 2007 Jun;17(3):238-45. doi: 10.1111/j.1600-0838.2006.00557.x. Epub 2006 Jun 15. PMID 16774652
- [Background] Ezzat AM, Whittaker JL, Brussoni M, Masse L, Emery CA. Translation and cross-cultural adaptation of the English version of the knee self-efficacy scale. Clinical journal of Sport Medicine. 2019;29(3):e57-58.
- [Background] Miller RP, Kori S, Todd D. The Tampa Scale: a measure of kinesiophobia. Clinical Journal of Pain. 1991;7(1):51-52.
- [Background] Kvist J, Ek A, Sporrstedt K, Good L. Fear of re-injury: a hindrance for returning to sports after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2005 Jul;13(5):393-7. doi: 10.1007/s00167-004-0591-8. Epub 2005 Feb 10. PMID 15703963
- [Background] Undheim MB, Cosgrave C, King E, Strike S, Marshall B, Falvey E, Franklyn-Miller A. Isokinetic muscle strength and readiness to return to sport following anterior cruciate ligament reconstruction: is there an association? A systematic review and a protocol recommendation. Br J Sports Med. 2015 Oct;49(20):1305-10. doi: 10.1136/bjsports-2014-093962. Epub 2015 Jun 23. PMID 26105017
- [Background] Amireault S, Godin G. The Godin-Shephard leisure-time physical activity questionnaire: validity evidence supporting its use for classifying healthy adults into active and insufficiently active categories. Percept Mot Skills. 2015 Apr;120(2):604-22. doi: 10.2466/03.27.PMS.120v19x7. Epub 2015 Mar 23. PMID 25799030
- [Background] Toomey CM, Whittaker JL, Nettel-Aguirre A, Reimer RA, Woodhouse LJ, Ghali B, Doyle-Baker PK, Emery CA. Higher Fat Mass Is Associated With a History of Knee Injury in Youth Sport. J Orthop Sports Phys Ther. 2017 Feb;47(2):80-87. doi: 10.2519/jospt.2017.7101. PMID 28142363
- [Background] Cleveland RJ, Alvarez C, Schwartz TA, Losina E, Renner JB, Jordan JM, Callahan LF. The impact of painful knee osteoarthritis on mortality: a community-based cohort study with over 24 years of follow-up. Osteoarthritis Cartilage. 2019 Apr;27(4):593-602. doi: 10.1016/j.joca.2018.12.008. Epub 2018 Dec 22. PMID 30583096
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Talma H, Chinapaw MJ, Bakker B, HiraSing RA, Terwee CB, Altenburg TM. Bioelectrical impedance analysis to estimate body composition in children and adolescents: a systematic review and evidence appraisal of validity, responsiveness, reliability and measurement error. Obes Rev. 2013 Nov;14(11):895-905. doi: 10.1111/obr.12061. Epub 2013 Jul 12. PMID 23848977
- [Background] Leahy S, O'Neill C, Sohun R, Jakeman P. A comparison of dual energy X-ray absorptiometry and bioelectrical impedance analysis to measure total and segmental body composition in healthy young adults. Eur J Appl Physiol. 2012 Feb;112(2):589-95. doi: 10.1007/s00421-011-2010-4. Epub 2011 May 26. PMID 21614505
- [Background] Roos EM, Dahlberg L. Positive effects of moderate exercise on glycosaminoglycan content in knee cartilage: a four-month, randomized, controlled trial in patients at risk of osteoarthritis. Arthritis Rheum. 2005 Nov;52(11):3507-14. doi: 10.1002/art.21415. PMID 16258919
- [Background] Munukka M, Waller B, Hakkinen A, Nieminen MT, Lammentausta E, Kujala UM, Paloneva J, Kautiainen H, Kiviranta I, Heinonen A. Physical Activity Is Related with Cartilage Quality in Women with Knee Osteoarthritis. Med Sci Sports Exerc. 2017 Jul;49(7):1323-1330. doi: 10.1249/MSS.0000000000001238. PMID 28240703
- [Background] Koli J, Multanen J, Kujala UM, Hakkinen A, Nieminen MT, Kautiainen H, Lammentausta E, Jamsa T, Ahola R, Selanne H, Kiviranta I, Heinonen A. Effects of Exercise on Patellar Cartilage in Women with Mild Knee Osteoarthritis. Med Sci Sports Exerc. 2015 Sep;47(9):1767-74. doi: 10.1249/MSS.0000000000000629. PMID 25668399
- [Background] Guermazi A, Alizai H, Crema MD, Trattnig S, Regatte RR, Roemer FW. Compositional MRI techniques for evaluation of cartilage degeneration in osteoarthritis. Osteoarthritis Cartilage. 2015 Oct;23(10):1639-53. doi: 10.1016/j.joca.2015.05.026. Epub 2015 Jun 5. PMID 26050864
- [Background] Matzat SJ, van Tiel J, Gold GE, Oei EH. Quantitative MRI techniques of cartilage composition. Quant Imaging Med Surg. 2013 Jun;3(3):162-74. doi: 10.3978/j.issn.2223-4292.2013.06.04. PMID 23833729
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Conner-Spady BL, Marshall DA, Bohm E, Dunbar MJ, Loucks L, Al Khudairy A, Noseworthy TW. Reliability and validity of the EQ-5D-5L compared to the EQ-5D-3L in patients with osteoarthritis referred for hip and knee replacement. Qual Life Res. 2015 Jul;24(7):1775-84. doi: 10.1007/s11136-014-0910-6. Epub 2015 Jan 3. PMID 25555837
- [Background] Bilbao A, Garcia-Perez L, Arenaza JC, Garcia I, Ariza-Cardiel G, Trujillo-Martin E, Forjaz MJ, Martin-Fernandez J. Psychometric properties of the EQ-5D-5L in patients with hip or knee osteoarthritis: reliability, validity and responsiveness. Qual Life Res. 2018 Nov;27(11):2897-2908. doi: 10.1007/s11136-018-1929-x. Epub 2018 Jul 5. PMID 29978346
- [Background] Kersten P, White PJ, Tennant A. The consultation and relational empathy measure: an investigation of its scaling structure. Disabil Rehabil. 2012;34(6):503-9. doi: 10.3109/09638288.2011.610493. Epub 2011 Oct 8. PMID 21981037
- [Background] Mercer SW, Maxwell M, Heaney D, Watt GC. The consultation and relational empathy (CARE) measure: development and preliminary validation and reliability of an empathy-based consultation process measure. Fam Pract. 2004 Dec;21(6):699-705. doi: 10.1093/fampra/cmh621. Epub 2004 Nov 4. PMID 15528286
- [Derived] Whittaker JL, Cammalleri A, Archibald C, Brooks-Hill A, Chin P, Clark S, Davis JC, Hoens AM, Hunt MA, Kausky K, Ko A, Leveille L, Li LC, Lodhia P, Losciale JM, Miciak M, Mosewich AD, Sheikh A, Silvester-Lee T, Truong LK, Wade D, Wilson DR, Xie H, Yan XH, Roos EM. Digital education and exercise therapy versus minimal intervention for young people at high risk of early onset knee osteoarthritis after ACL reconstruction: a study protocol for the Stop OsteoARthritis (SOAR) randomized controlled trial. Trials. 2025 Jun 20;26(1):213. doi: 10.1186/s13063-025-08896-6. PMID 40542399